CLINICAL TRIAL: NCT01236612
Title: Experimental Human Malaria Infection After Immunization With Plasmodium Falciparum Sporozoites Under Chloroquine Prophylaxis
Acronym: EHMI9
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EHMI9
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Plasmodium; falciparum; malaria; chloroquine; immunity
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Immunization; Proguanil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Immunization + bloodstage challenge (Experimental)
  Interventions: Drug: Chloroquine prophylaxis; Biological: Immunization; Biological: Plasmodium falciparum Bloodstage challenge; Drug: Malarone treatment
- Immunization + mosquito challenge (Active Comparator)
  Interventions: Drug: Chloroquine prophylaxis; Biological: Immunization; Biological: Plasmodium falciparum mosquito challenge; Drug: Malarone treatment
- Control - Bloodstage challenge (Placebo Comparator)
  Interventions: Biological: Plasmodium falciparum Bloodstage challenge; Drug: Malarone treatment
- Control - Mosquito challenge (Placebo Comparator)
  Interventions: Biological: Plasmodium falciparum mosquito challenge; Drug: Malarone treatment

INTERVENTIONS:
Drug: Chloroquine prophylaxis — The chloroquine dose used will be 300mg for the first two days, followed by 300mg per week, for 13 weeks.
  Arms: Immunization + bloodstage challenge; Immunization + mosquito challenge
Biological: Immunization — Groups 1 and 2 will be immunized with 3 times 15 bites of Pf infected mosquitoes under chloroquine prophylaxis.
  Arms: Immunization + bloodstage challenge; Immunization + mosquito challenge
Biological: Plasmodium falciparum Bloodstage challenge — Groups 1 and 3 will be challenged by intravenous administration of Plasmodium falciparum infected erythrocytes.
  Arms: Control - Bloodstage challenge; Immunization + bloodstage challenge
Biological: Plasmodium falciparum mosquito challenge — Groups 2 and 4 will be challenged by the bites of 5 Plasmodium falciparum infected mosquitoes.
  Arms: Control - Mosquito challenge; Immunization + mosquito challenge
Drug: Malarone treatment — When thick smear positive, of ar day 21 after challenge, all volunteers will be treated with malarone.
  Other Names: atovaquon/proguanil

SUMMARY:
Malaria is one of the major infectious diseases in the world with a tremendous impact on the quality of life significantly contributing to the ongoing poverty in endemic countries. It causes almost one million deaths per year, the majority of which are children under the age of five. The malaria parasite enters the human body through the skin, by the bite of an infected mosquito. Subsequently, it invades the liver and develops and multiplies inside the hepatocytes. After a week, the hepatocytes burst open and the parasites are released in the blood stream, causing the clinical phase of the disease.

As a unique opportunity to study malaria immunology and efficacy of immunisation strategies, a protocol has been developed in the past to conduct experimental human malaria infections (EHMIs). EHMIs generally involve small groups of malaria-naïve volunteers infected via the bites of P. falciparum infected laboratory-reared Anopheline mosquitoes. Although potentially serious or even lethal, Plasmodium falciparum (P.falciparum) malaria can be radically cured at the earliest stages of blood infection where risks of complications are virtually absent.

The investigators have shown previously, that healthy human volunteers can be protected from a malaria mosquito challenge by immunization with mosquito-bites under chloroquine prophylaxis (CPS immunization). However, it is unknown whether this protection is based on immunity directed towards the liver- or the blood stage of the disease. For future development of vaccines and understanding of protective immunity to malaria, it is important to investigate at which level protective immunity is generated by CPS immunization. Therefore, we aim to investigate whether CPS immunization confers protection to a blood-stage challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and < 35 years healthy volunteers (males or females)
2. Good health based on history and clinical examination
3. Negative pregnancy test
4. Use of adequate contraception for females
5. All volunteers must sign the informed consent form demonstrating their understanding of the meaning and procedures of the study
6. Volunteer agrees to inform the general practitioner and agrees to sign a request to release medical information concerning contra-indications for participation in the study
7. Willingness to undergo a Pf mosquito or blood stage challenge
8. For volunteers not living in Nijmegen: agreement to stay in a hotel room close to the trial center during a part of the study (for groups 1 and 3 from challenge day till 3 days after treatment, for groups 2 and 4 from 5 days after challenge till 3 days after treatment)
9. Reachable (24/7) by mobile phone during the whole study period
10. Living with a third party that could contact the clinicians in case of alteration of consciousness or agreement to stay in a hotel room close to the trial center during a part of the study (for groups 1 and 3 from challenge day till 3 days after treatment, for groups 2 and 4 from 5 days after challenge till 3 days after treatment)
11. Available to attend all study visits
12. Agreement to refrain from blood donation to Sanquin or for other purposes, during the study period until 393
13. Willingness to undergo HIV, hepatitis B and hepatitis C tests
14. Negative urine toxicology screening test at screening visit and day before challenge
15. Willingness to take a prophylactic regime of chloroquine and curative regimen of Malarone®

Exclusion Criteria:

1. History of malaria
2. Plans to travel to malaria endemic areas during the study period
3. Plans to travel outside of the Netherlands during the challenge period
4. Previous participation in any malaria vaccine study and/or positive serology for Pf
5. Symptoms, physical signs and laboratory values suggestive of systemic disorders including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric, and other conditions which could interfere with the interpretation of the study results or compromise the health of the volunteers
6. History of diabetes mellitus or cancer (except basal cell carcinoma of the skin)
7. History of arrhythmias or prolonged QT-interval
8. Positive family history in 1st and 2nd degree relatives for cardiac disease < 50 years old
9. An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system
10. Clinically significant abnormalities in electrocardiogram (ECG) at screening
11. Body Mass Index (BMI) below 18 or above 30 kg/m2
12. Any clinically significant deviation from the normal range in biochemistry or hematology blood tests or in urine analysis
13. Positive HIV, HBV or HCV tests
14. Participation in any other clinical study within 30 days prior to the onset of the study
15. Enrollment in any other clinical study during the study period
16. Pregnant or lactating women
17. Volunteers unable to give written informed consent
18. Volunteers unable to be closely followed for social, geographic or psychological reasons
19. Previous history of drug or alcohol abuse interfering with normal social function during a period of one year prior to enrolment in the study
20. A history of psychiatric disease
21. Known hypersensitivity to anti-malaria drugs
22. The use of chronic immunosuppressive drugs, antibiotics, or other immune modifying drugs within three months of study onset (inhaled and topical corticosteroids are allowed) and during the study period
23. Contra-indications to Malarone® or chloroquine including treatment taken by the volunteer that interferes with Malarone® or chloroquine
24. Any confirmed or suspected immunosuppressive or immunodeficient condition, including asplenia
25. Co-workers of the departments of Medical Microbiology or Internal Medicine of the RUNMC
26. A history of sickle cell anemia, sickle cell trait, thalassemia, thalassemia trait or G6PD deficiency

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Duration of prepatent period as measured by microscopy | 21 days after challenge
Parasitemia and kinetics of parasitemia as measured by PCR | 21 days after challenge
Frequency of signs or symptoms in study groups | 21 days after challenge

SECONDARY OUTCOMES:
Antibody production in groups 1, 2, 3 and 4 | 393 days
Cellular immune response in groups 1, 2, 3 and 4 | 393 days
Cytokine profile in groups 1, 2, 3 and 4 | 393 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Sauerwein, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Background] Roestenberg M, McCall M, Hopman J, Wiersma J, Luty AJ, van Gemert GJ, van de Vegte-Bolmer M, van Schaijk B, Teelen K, Arens T, Spaarman L, de Mast Q, Roeffen W, Snounou G, Renia L, van der Ven A, Hermsen CC, Sauerwein R. Protection against a malaria challenge by sporozoite inoculation. N Engl J Med. 2009 Jul 30;361(5):468-77. doi: 10.1056/NEJMoa0805832. PMID 19641203
- [Result] Bijker EM, Bastiaens GJ, Teirlinck AC, van Gemert GJ, Graumans W, van de Vegte-Bolmer M, Siebelink-Stoter R, Arens T, Teelen K, Nahrendorf W, Remarque EJ, Roeffen W, Jansens A, Zimmerman D, Vos M, van Schaijk BC, Wiersma J, van der Ven AJ, de Mast Q, van Lieshout L, Verweij JJ, Hermsen CC, Scholzen A, Sauerwein RW. Protection against malaria after immunization by chloroquine prophylaxis and sporozoites is mediated by preerythrocytic immunity. Proc Natl Acad Sci U S A. 2013 May 7;110(19):7862-7. doi: 10.1073/pnas.1220360110. Epub 2013 Apr 18. PMID 23599283
- [Derived] Coffeng LE, Hermsen CC, Sauerwein RW, de Vlas SJ. The Power of Malaria Vaccine Trials Using Controlled Human Malaria Infection. PLoS Comput Biol. 2017 Jan 12;13(1):e1005255. doi: 10.1371/journal.pcbi.1005255. eCollection 2017 Jan. PMID 28081133
- [Derived] Nahrendorf W, Scholzen A, Bijker EM, Teirlinck AC, Bastiaens GJ, Schats R, Hermsen CC, Visser LG, Langhorne J, Sauerwein RW. Memory B-cell and antibody responses induced by Plasmodium falciparum sporozoite immunization. J Infect Dis. 2014 Dec 15;210(12):1981-90. doi: 10.1093/infdis/jiu354. Epub 2014 Jun 25. PMID 24970846